CLINICAL TRIAL: NCT00383955
Title: Comparison of Screening Tools for Coronary Artery Disease With Thallium Scintigraphy in Adult Population in Karachi.
Brief Title: Comparison of Screening Tools for Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Wellcome Trust (Other)
Other Study IDs: 078440/Z/05/Z
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2006-10

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Coronary artery disease (CAD) is a silent killer that may go undetected for years. It is the leading cause of death with no limitation to geographic boundaries accounting to about 16.7 million deaths world wide. Different studies have shown that South Asians populations are more prone to CAD where it is emerging as an epidemic. According to a study conducted in Karachi it is estimated that the overall prevalence of cardiovascular diseases in Pakistan is 26.9% with 23.7% in men and 30.0% in women. However tools for measuring CAD have not being adequately validated. This study is designed to develop screening tools and to determine test characteristics of Rose Questionnaire and Minnesota Coded ECG alone and in combination for diagnosis of CAD, using MPI as gold standard in Pakistan.

DETAILED DESCRIPTION:
Design: The proposed study is a cross sectional study of a population sample of 450 subjects aged > 40 years, and stratified by gender, residing in 12 randomly selected communities in Karachi, Pakistan.

The target population for this study would be drawn from an existing population based study entitled "Population based strategies for effective control of high blood pressure in Pakistan" (parent study), conducted by the primary supervisor and study director (TJ) in Karachi Subjects aged > 40 years would be eligible. Detailed information on each participant would be obtained from data collected for the parent study. This includes a) socio-demographic characteristics such as level of education, occupation, economic status, ethnicity, tobacco use , physical activity defined on the basis of International Physical Activity Questionnaire, dietary habits (food frequency questionnaire), family history of CAD, and the WHO standard Rose questionnaire (RQ) for coronary artery disease (CAD) (b) anthropometry including height, weight, waist and hip circumference (c) laboratory tests including fasting blood glucose, lipid profile, serum creatinine, and urine albumin to creatinine ratio. The community health workers (CHW) would administer RQ and obtain 12-lead EKG. They would give an appointment to subjects for MPI at the Aga Khan University Hospital. Each individual will then go through an exercise treadmill test (symptom limited Bruce or modified Bruce protocols) if able to walk, or pharmacological stress by the infusion of dobutamine or dipyridamole if unable to walk. The results of MPI study would be delivered to the subjects with interpretation by cardiologists, and referral to a physician (as appropriate).

Classification of Screening instruments: ECG will be Minnesota coded by two trained and independent coders, and discrepant reports will be resolved with a third independent coder. All cases of probable or possible CAD on Minnesota coding of ECG would be classified as "MC ECG positive for CAD" RQ will be coded according to standardized criteria into "positives for "angina" and "history of possible infarction" . Presence of either one would be classified as "RQ positive for CAD".

ELIGIBILITY:
Inclusion Criteria:

1. Adult resident of Karachi residing in selected clusters
2. Age > 40 years

Exclusion Criteria:

1. Clinical Heart Failure
2. Severe Disease e.g. Cancer
3. Pregnant or lactating women
4. People with limited mobility
5. People not willing to participate

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tazeen H Jafar, MD, MPH, Study Director — Aga Khan University; Dr. Shazia S Abbas, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Hospital, Karachi, Sindh, Pakistan